CLINICAL TRIAL: NCT05276050
Title: Circuitry-Guided Smoking Cessation in Schizophrenia (UH3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-23-0632; UH3DA047685 (NIH)
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Nicotine Addiction; Schizophrenia
Keywords: Transcranial magnetic stimulation; schizophrenia; smoking; nicotine; tobacco
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Schizophrenia; Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study group (Experimental): Participants in this group will receive active F8-coil delivered rTMS.
  Interventions: Device: active F8-coil delivered rTMS
- Active control group (Active Comparator): Participants in this group will receive active H-coil delivered rTMS.
  Interventions: Device: active H-coil delivered rTMS

INTERVENTIONS:
Device: active F8-coil delivered rTMS — Multiple trains of rTMS in a day, for multiple days.
  Arms: Study group
Device: active H-coil delivered rTMS — Multiple trains of rTMS in a day, for multiple days.
  Arms: Active control group

SUMMARY:
Patients with schizophrenia spectrum disorder (SSD) will be exposed to active repetitive transcranial magnetic stimulation (rTMS) from F8 coil or active rTMS from H coil for smoking cessation. Smoking and brain functional connectivity changes will be assessed at baseline, different stages of rTMS and/or follow-ups.

DETAILED DESCRIPTION:
Neuroimaging studies suggest that high rate of smoking in patients with schizophrenia may be due to an overlap of nicotine addiction-related circuitries and schizophrenia-related circuitries, such that schizophrenia impacts some of the same circuitries that increase risks for severe nicotine addiction in general. Those identified overlapping circuitries have been linked to several key features of nicotine addiction and can be represented by resting-state functional connectivities. The investigators aim to develop a TMS method targeting special brain circuits that are both smoking cessation and schizophrenia-related. If the corresponding brain circuits were successfully modulated, the treatment efficacy will be significantly improved and schizophrenia patients will benefit from the TMS treatment of smoking cessation.

The F8 coil based rTMS is not FDA approved for smoking cessation at this point, the rTMS with H4 coil is FDA-cleared for short-term smoking cessation in the general population, its efficacy in SSD has not been evaluated. In this protocol, the investigators will compare them in patients with schizophrenia spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between ages 22-65 years
2. Ability to give written informed consent
3. Smoking in the last one year or more and average cigarette per day ≥ 5 in the past 4 weeks
4. Diagnosed with schizophrenia-spectrum disorder and Evaluation to Sign Consent (ESC) above10.
5. Is currently under the care of a licensed primary care provider or mental healthcare provider (e.g., psychiatrist, psychologist, nurse practitioner, licensed clinical social worker).
6. Agrees to: (a) provide written permission, as requested, to allow any and all forms of communication between the investigators and study staff and any health care provider who currently provides and/or has provided service to the subject within two years of study enrollment; and (b) provide the names and verifiable contact information (name, email and mailing address, mobile and land-line phone number, as applicable) of at least two reliable persons ≥ age 22, who reside within a 30-minute drive of the subject's residence, and whom the research staff is at liberty to contact, as deemed necessary, for the duration of study participation.

Exclusion Criteria:

1. Persons with a first-degree relative with inherited epilepsy, seizure disorder, or seizures or persons who answer "yes" to any of the parts (A. - G.) of Question 3 of an epilepsy screening questionnaire.
2. Had smoking cessation treatment, clinical trial, or nicotine replacements within the past four weeks.
3. Significant alcohol or other drug use (substance dependence within 6 months or substance abuse within 1 month) other than nicotine or marijuana dependence.
4. Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, CNS infection or tumor, other significant brain neurological conditions.
5. Taking > 400 mg clozapine/day or Failed TMS screening questionnaire.
6. Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
7. History of head injury with loss of consciousness over 10 minutes; history of brain surgery
8. Cannot refrain from using alcohol and/or marijuana 24 hours or more & cigarette smoking one hour or more prior to experiments.
9. Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive pregnancy test) or has had unprotected sexual intercourse without birth control in the last 4 weeks.
10. Moderate-High Risk of suicide according to the Columbia - Suicide Severity Rating Scale (C- SSRS) Screen Version - Recent (i.e. answers YES to Question 3 and NO to Question 6 (Moderate risk); or answers YES to Questions 4, 5, or 6 (High risk) or in the clinical judgement of the investigator or the study psychiatrist.
11. In the medical opinion of the investigator, subjects with the following circumstances or conditions which can increase the risk of seizures may be excluded: sleep deprivation; major depressive disorder comorbid with dementia, underweight status; concurrent use of cephalosporins and antiarrhythmics (particularly propranolol); metabolic abnormalities (hyponatremia, hypocalcemia, hypomagnesemia, hypoglycemia, hyperglycemia, renal failure/uremia, liver failure); raised blood concentrations of proconvulsant medications due to reduced clearance (e.g. secondary to initiation of antibiotics for treatment of infections); alcohol withdrawal; use of stimulants, such as cocaine or MDMA; use of immunosuppressive therapy with cyclosporine, tacrolimus and other agents that can cause the posterior reversible leukoencephalopathy syndrome; dialysis; systemic infection, and fever itself.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Resting-state functional connectivity (rsFC) from functional magnetic resonance imaging (fMRI) | 1 month
  The strength of rsFC from fMRI is used to represent the brain activities that are corresponding to the TMS effect on smoking reduction/cessation.
Cigarette per day | 1 month
  Cigarette per day (CPD) is measured to index smoking reduction and cessation.

SECONDARY OUTCOMES:
Fagerstrom Test for Nicotine Dependence (FTND) | 1 month
  Fagerstrom Test for Nicotine Dependence (FTND) represents the severity of nicotine severity.
nicotine/creatinine | 1 month
  nicotine/creatinine is a index of smoking status.
End-expired carbon monoxide (CO) | 1 month
  End-expired CO measure is an instant measure of smoking status.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No